CLINICAL TRIAL: NCT04203576
Title: First In Human Clinical Investigation of the FIRE1 System in Heart Failure Patients
Brief Title: First in Human Clinical Investigation of the FIRE1 System in Heart Failure Patients (FUTURE-HF)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundry Innovation & Research 1, Limited (FIRE1) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF01-CID04
Record Dates: First submitted 2019-12-12; First posted 2019-12-18 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Cardiovascular Disease
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FIRE1 System (Experimental): FIRE1 System
  Interventions: Device: FIRE1 System

INTERVENTIONS:
Device: FIRE1 System — FIRE1 System

SUMMARY:
First in Human Clinical Investigation of the FIRE1 Device/System to evaluate the feasibility and safety of implanting the FIRE1 system in up to 50 stable HF patients.

DETAILED DESCRIPTION:
Eligible patients who have HF and were hospitalised/treated for an episode of worsening HF within the last 6 months. This non-randomised FIH trial will enrol a total of 50 patients and the primary safety and technical endpoints will be assessed at 3 months. Safety measures will include an assessment of all adverse events. Subjects will remain in this study for 24 months.

ELIGIBILITY:
Main Inclusion Criteria

* Adults 18 years or older with heart failure with any of the following in the past 6 months: a decompensation due to heart failure resulting in a heart failure hospitalisation, heart failure treatment in a hospital day-care setting or urgent outpatient heart failure visit
* Receiving treatment in accordance with internationally recognised guidelines.
* Signed patient informed consent form

Main Exclusion Criteria:

* Significant comorbidity that would interfere with the ability to safely complete the clinical investigation protocol
* Patients with an estimated Glomerular Filtration Rate (eGFR) < 30 ml/min
* Patients with IVC filter placement in situ, abnormal IVC or femoral venous anatomy or known congenital malformation or absence of IVC or occlusive or free-floating thrombus in the IVC
* Patients with implantable ventricular assist device (LVAD, RVAD, BiVAD) in situ
* Patients with Cardiovascular Implantable Electronic Device (CIED) implanted ≤ 3 months prior to enrolment
* Patients with conditions associated with occlusion of the IVC, iliac or common femoral veins (e.g. venous leg ulcers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Procedural success and freedom from FIRE1 sensor complications | 3 months
  The primary, composite endpoint is success of the FIRE1 sensor, which includes procedural success defined as sensor deployment at the intended site without acute device or procedural related complications and freedom from sensor complications including device migration, clinically significant fracture and/ or clinically significant perforation of the Inferior Vena Cava (IVC) or symptomatic caval thrombosis.
Primary Technical Endpoint - Signal acquisition from the FIRE1 sensor | 3 months
  Technical success defined as signal acquisition immediately post implantation and at an attended clinic visit.

SECONDARY OUTCOMES:
Secondary Safety Endpoint: Freedom from symptomatic access site thrombosis confirmed by ultrasound | 3 months
  Freedom from symptomatic access site thrombosis confirmed by ultrasound. Freedom from a significant hematoma (defined as requiring intervention, transfusion or prolonging hospitalisation).
Secondary Technical Endpoint - Successful transmission of FIRE1 signal. | 3 months
  Successful transmission of a FIRE1 sensor reading from the patient's home.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Kent, Study Director — Clinical Director
Locations (13):
- Czechia (2):
  - Nemocnice Na Homolce, Prague, Praha 5
  - Fakultní Nemocnice Brno, Brno
- Georgia (2):
  - Israeli-Georgian Medical Research Clinic Helsikor, Tbilisi
  - Tbilisi Heart and Vascular Clinic, Tbilisi
- Galway University Hospital, Galway, Ireland
- Netherlands (2):
  - Erasmus University Medical Center, Rotterdam, Dr. Molewaterplein 40
  - University Medical Center, Groningen, Groningen, Hanzeplein 1
- United Kingdom (6):
  - Royal Bournemouth Hospital, Bournemouth
  - Golden Jubilee National Hospital, Glasgow
  - Glenfield Hospital, Leicester
  - Royal Brompton Hospital Sydney Street, London
  - Queen Alexandra Hospital, Portsmouth
  - University Hospital Southampton, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalra PR, Gogorishvili I, Khabeishvili G, Malek F, Toman O, Critoph C, Flett AS, Cowburn PJ, Mehra MR, Sheridan WS, Britton JR, Buxo T, Kealy RM, Kent A, Greene BR, Guha K, Gardner RS, Loke I, Vazir A, Brugts JJ, Gray A, Testani JM, Damman K. First-in-Human Implantable Inferior Vena Cava Sensor for Remote Care in Heart Failure: FUTURE-HF. JACC Heart Fail. 2025 Jun;13(6):1000-1010. doi: 10.1016/j.jchf.2025.01.019. Epub 2025 Apr 9. PMID 40208140